CLINICAL TRIAL: NCT00073515
Title: A Phase 2, Multicenter, Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of Alfimeprase for Restoring Function in Occluded Central Venous Catheters
Brief Title: Trial of a Novel Fibrinolytic (Alfimeprase) to Clear Thrombosed Vascular Access Devices
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ARCA Biopharma, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: HA003; NuCath-1
Record Dates: First submitted 2003-11-21; First posted 2003-11-25 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2005-06

CONDITIONS: Catheters, Indwelling
Keywords: central venous access device; thrombosis; central venous catheter; thrombolysis; fibrinolysis
MeSH Terms: conditions — Thrombosis | interventions — alfimeprase

INTERVENTIONS:
Drug: Alfimeprase

SUMMARY:
This trial is for patients with a central venous catheter (a vascular access device) that is not functioning properly (unable to withdraw blood). The trial compares a new blood clot dissolving agent (alfimeprase) against the currently used treatment.

ELIGIBILITY:
Subjects must:

* have a dysfunctional Central Venous Access Device (CVAD) defined as unable to withdraw 3 mL blood
* have had the device in place for > 48 hours
* be clinically stable
* be 18 or older
* give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States